CLINICAL TRIAL: NCT05318144
Title: Prognostic Value of Serum Melatonin as a Biomarker for the Determination of Severe COVID-19 Infection in Pregnant Women
Brief Title: Melatonin Levels on COVID-19 Positive Pregnant Women
Status: Completed | Type: Observational
Sponsor: Nazan Yurtcu MD (Other)
Responsible Party: Sponsor-Investigator, Nazan Yurtcu MD, Assistant Professor, Cumhuriyet University
Organization: Cumhuriyet University (Other)
Other Study IDs: COVID-19 and pregnancy
Record Dates: First submitted 2022-04-06; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Pregnancy Related; Pregnancy Complications
Keywords: COVID-19; SARS-CoV-2; Melatonine; pregnancy; pregnancy outcomes
MeSH Terms: conditions — Pregnancy Complications; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PCR (-) symptomatic: control group, pregnant women with negative COVID-19 Polymerase Chain Reaction (PCR) test
- PCR (+) asymptomatic: Pregnant women who have a positive COVID-19 PCR test and have had the infection without symptoms
- PCR (+) mild-moderate: Pregnant women with positive COVID-19 PCR test and mild to moderate symptoms and inpatient treatment
- PCR (+) severe COVID-19: Pregnant women with positive COVID-19 PCR test and severe symptoms

INTERVENTIONS:
Other:

SUMMARY:
This study aimed to investigate the prognostic value of serum melatonin as a biomarker for the determination of severe COVID-19 infection in pregnant women.

Four study groups were formed, including pregnant women with a positive COVID-19 PCR test, severe symptoms, and inpatient treatment. Pregnant women who had complaints similar to COVID-19 infection or had no complaints, but had a PCR test due to the surveillance program and negative test results were included in the control group.

Methods and Main Outcome measure: Laboratory values of the cases at the time of diagnosis parameters were collected.

Melatonin levels decrease in pregnant women with COVID-19 symptoms, the severity of symptoms increases. In addition, patients with low melatonin levels have an increase in infection parameters and an increase in the hospital stay.

DETAILED DESCRIPTION:
A total of 228 pregnant women included in this prospective controlled study between June 20021 and June 2022 at Gynecology and Obstetrics Department of Health Sciences University Samsun Training and Research Hospital.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with a positive COVID-19 PCR test and severe symptoms and inpatient treatment. Pregnant women who had complaints similar to COVID-19 infection or had no complaints but had a PCR test due to the surveillance program and negative test results were included in the control group. Pregnant women who had contact with people with COVID-19 infection and had a PCR test due to the surveillance program and had positive results, but no complaints were included in the other study group. The PCR test of pregnant women who had complaints and needed inpatient treatment during the COVID-19 infection was confirmed, and the COVID-19 infection was graded according to WHO's criteria. Pregnant women with viral infection with symptoms compatible with infection and virus isolation in any culture samples collected at admission were included in the patient group with PCR positive mild-moderate and severe COVID-19 infection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with COVID-19 and control groups
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Melatonin level | 6 year
  Melatonin level of pregnant women with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Oral, Study Chair — Halic University Faculty of Medicine, Department of Obstetrics and Gynecology
Locations (1):
- Samsun Training and Research Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
June 2021- December 2021

REFERENCES:
- [Background] Di Mascio D, Buca D, Berghella V, Khalil A, Rizzo G, Odibo A, Saccone G, Galindo A, Liberati M, D'Antonio F. Counseling in maternal-fetal medicine: SARS-CoV-2 infection in pregnancy. Ultrasound Obstet Gynecol. 2021 May;57(5):687-697. doi: 10.1002/uog.23628. PMID 33724545
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Huntley BJF, Huntley ES, Di Mascio D, Chen T, Berghella V, Chauhan SP. Rates of Maternal and Perinatal Mortality and Vertical Transmission in Pregnancies Complicated by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Co-V-2) Infection: A Systematic Review. Obstet Gynecol. 2020 Aug;136(2):303-312. doi: 10.1097/AOG.0000000000004010. PMID 32516273
- [Result] Yurtcu N, Caliskan C, Celik S. Serum Melatonin as a Biomarker for Assessment of Late-term and Postterm Pregnancies in Women without Spontaneous Onset of Labor. Z Geburtshilfe Neonatol. 2021 Dec;225(6):499-505. doi: 10.1055/a-1479-3220. Epub 2021 May 31. PMID 34058776
- [Result] Head Zauche L, Wallace B, Smoots AN, Olson CK, Oduyebo T, Kim SY, Peterson EE, Ju J, Beauregard J, Wilcox AJ, Rose CE, Meaney-Delman D, Ellington SR. Receipt of mRNA COVID-19 vaccines preconception and during pregnancy and risk of self-reported spontaneous abortions, CDC v-safe COVID-19 Vaccine Pregnancy Registry 2020-21. Res Sq [Preprint]. 2021 Aug 9:rs.3.rs-798175. doi: 10.21203/rs.3.rs-798175/v1. PMID 34401872
- [Result] Wastnedge EAN, Reynolds RM, van Boeckel SR, Stock SJ, Denison FC, Maybin JA, Critchley HOD. Pregnancy and COVID-19. Physiol Rev. 2021 Jan 1;101(1):303-318. doi: 10.1152/physrev.00024.2020. Epub 2020 Sep 24. PMID 32969772
- [Result] Wong SF, Chow KM, Leung TN, Ng WF, Ng TK, Shek CC, Ng PC, Lam PW, Ho LC, To WW, Lai ST, Yan WW, Tan PY. Pregnancy and perinatal outcomes of women with severe acute respiratory syndrome. Am J Obstet Gynecol. 2004 Jul;191(1):292-7. doi: 10.1016/j.ajog.2003.11.019. PMID 15295381
- [Result] Di Mascio D, Khalil A, Saccone G, Rizzo G, Buca D, Liberati M, Vecchiet J, Nappi L, Scambia G, Berghella V, D'Antonio F. Outcome of coronavirus spectrum infections (SARS, MERS, COVID-19) during pregnancy: a systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2020 May;2(2):100107. doi: 10.1016/j.ajogmf.2020.100107. Epub 2020 Mar 25. PMID 32292902
- [Result] Voiculescu SE, Zygouropoulos N, Zahiu CD, Zagrean AM. Role of melatonin in embryo fetal development. J Med Life. 2014 Oct-Dec;7(4):488-92. PMID 25713608
- [Result] Uzun M, Gencer M, Turkon H, Oztopuz RO, Demir U, Ovali MA. Effects of Melatonin on Blood Pressure, Oxidative Stress and Placental Expressions of TNFalpha, IL-6, VEGF and sFlt-1 in RUPP Rat Model of Preeclampsia. Arch Med Res. 2017 Oct;48(7):592-598. doi: 10.1016/j.arcmed.2017.08.007. Epub 2018 Feb 1. No abstract available. PMID 29397206
- [Result] Anderson G, Maes M, Markus RP, Rodriguez M. Ebola virus: melatonin as a readily available treatment option. J Med Virol. 2015 Apr;87(4):537-43. doi: 10.1002/jmv.24130. Epub 2015 Jan 21. PMID 25611054
- [Result] Anderson G, Reiter RJ. Melatonin: Roles in influenza, Covid-19, and other viral infections. Rev Med Virol. 2020 May;30(3):e2109. doi: 10.1002/rmv.2109. Epub 2020 Apr 21. PMID 32314850
- [Result] Nehme PA, Amaral FG, Middleton B, Lowden A, Marqueze E, Franca-Junior I, Antunes JLF, Cipolla-Neto J, Skene DJ, Moreno CRC. Melatonin profiles during the third trimester of pregnancy and health status in the offspring among day and night workers: A case series. Neurobiol Sleep Circadian Rhythms. 2019 Apr 13;6:70-76. doi: 10.1016/j.nbscr.2019.04.001. eCollection 2019 Jan. PMID 31236522
- [Result] Farnoosh G, Akbariqomi M, Badri T, Bagheri M, Izadi M, Saeedi-Boroujeni A, Rezaie E, Ghaleh HEG, Aghamollaei H, Fasihi-Ramandi M, Hassanpour K, Alishiri G. Efficacy of a Low Dose of Melatonin as an Adjunctive Therapy in Hospitalized Patients with COVID-19: A Randomized, Double-blind Clinical Trial. Arch Med Res. 2022 Jan;53(1):79-85. doi: 10.1016/j.arcmed.2021.06.006. Epub 2021 Jun 23. PMID 34229896
- [Result] Salles C. Correspondence COVID-19: Melatonin as a potential adjuvant treatment. Life Sci. 2020 Jul 15;253:117716. doi: 10.1016/j.lfs.2020.117716. Epub 2020 Apr 22. No abstract available. PMID 32334009
- [Result] Liset R, Gronli J, Henriksen RE, Henriksen TEG, Nilsen RM, Pallesen S. A randomized controlled trial on the effect of blue-blocking glasses compared to partial blue-blockers on melatonin profile among nulliparous women in third trimester of the pregnancy. Neurobiol Sleep Circadian Rhythms. 2021 Dec 29;12:100074. doi: 10.1016/j.nbscr.2021.100074. eCollection 2022 May. PMID 35024497